CLINICAL TRIAL: NCT00518466
Title: A Phase Ib, Open Label, Parallel-Design Single- and Multiple-Dose Study Comparing Modified Release Topiramate Formulations to Immediate Release Formulations of Topiramate Dosed in Combination With Immediate Release Phentermine in Obese Adults
Brief Title: Pharmacokinetic Comparison of Multiple Formulations of Topiramate and Phentermine in Obese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical, Vivus, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OB-102 / AA42851
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Topiramate; Phentermine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- treatment 1 (Experimental): One 7.5 mg phentermine hydrochloride IR capsule and two 25 mg topiramate MR capsules at Hour 0 on Day 1 of Period 1.
  One 7.5 mg phentermine hydrochloride IR capsule and one 25 mg topiramate MR capsule at Hour 0 on Days 1, 2, and 3 of Period 2.
  One 7.5 mg phentermine hydrochloride IR capsule and two 25 mg topiramate MR capsules at Hour 0 on Days 4 - 21 of Period 2.
  Interventions: Drug: topiramate; Drug: phentermine
- treatment 2 (Experimental): Two 7.5 mg phentermine hydrochloride IR capsules and four 25 mg topiramate MR capsules at Hour 0 on Day 1 of Period 1.
  One 7.5 mg phentermine hydrochloride IR capsule and one 25 mg topiramate MR capsule at Hour 0 on Days 1, 2, and 3 of Period 2.
  One 7.5 mg phentermine hydrochloride IR capsules and two 25 mg topiramate MR capsules at Hour 0 on Days 4, 5, and 6 of Period 2.
  Two 7.5 mg phentermine hydrochloride IR capsules (Cardinal) and three 25 mg topiramate MR capsules at Hour 0 on Days 7, 8, and 9 of Period 2.
  Two 7.5 mg phentermine hydrochloride IR capsules and four 25 mg topiramate MR capsules at Hour 0 on Days 10 - 21 of Period 2.
  Interventions: Drug: topiramate; Drug: phentermine
- treatment 3 (Experimental): Two 7.5 mg phentermine hydrochloride IR capsules and four 25 mg topiramate MR capsules at Hour 0 on Day 1 of Period 1.
  One 7.5 mg phentermine hydrochloride IR capsule and one 25 mg topiramate MR capsule at Hour 0 on Days 1, 2, and 3 of Period 2.
  Two 7.5 mg phentermine hydrochloride IR capsules and two 25 mg topiramate MR capsule at Hour 0 on Days 4, 5, and 6 of Period 2.
  Two 7.5 mg phentermine hydrochloride IR capsules and three 25 mg topiramate MR capsules at Hour 0 on Days 7, 8, and 9 of Period 2.
  Two 7.5 mg phentermine hydrochloride IR capsules and four 25 mg topiramate MR capsules at Hour 0 on Days 10 - 21 of Period 2.
  Interventions: Drug: topiramate; Drug: phentermine
- treatment 4 (Experimental): Half of a 37.5 mg phentermine hydrochloride IR tablet and one 100 mg topiramate IR tablet at Hour 0 on Day 1 of Period 1.
  One 7.5 mg phentermine hydrochloride IR capsule and one 25 mg topiramate IR tablet at Hour 0 on Days 1, 2, and 3 of Period 2.
  Half of a 37.5 mg phentermine hydrochloride IR tablet and two 25 mg topiramate IR tablets at Hour 0 on Days 4, 5, and 6 of Period 2.
  Half of a 37.5 mg phentermine hydrochloride IR tablet and three 25 mg topiramate IR tablets at Hour 0 on Days 7, 8, and 9 of Period 2.
  Half of a 37.5 mg phentermine hydrochloride IR tablet and one 100 mg topiramate IR tablet at Hour 0 on Days 10 - 21 of Period 2.
  Interventions: Drug: topiramate; Drug: phentermine

INTERVENTIONS:
Drug: topiramate — 25 mg modified-release capsules
  Arms: treatment 1; treatment 2; treatment 3
Drug: phentermine — 7.5 mg immediate-release capsules
  Arms: treatment 1; treatment 2; treatment 3
Drug: topiramate — 100 and 25 mg immediate-release tablets
  Arms: treatment 4
Drug: phentermine — 37.5 and 7.5 mg immediate-release tablets
  Arms: treatment 4

SUMMARY:
The primary objective of this study is to describe the single- and multiple-dose pharmacokinetic profiles of two novel formulations of topiramate and commercially available immediate release topiramate, all dosed with immediate release phentermine.

ELIGIBILITY:
Inclusion Criteria:

* Obese adults
* Body mass index between 30.0 and 42.0 kg/m2 (inclusive)
* Medically healthy with no clinically significant results of screening exams

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* History of glaucoma or increased intraocular pressure
* History of kidney stones
* Cholelithiasis or cholecystitis within 6 months
* Cardiovascular event within 6 months
* Obesity of known genetic or endocrine origin
* Recent weight instability
* Use of Very Low Calorie diet or participation in organized weight loss program within 3 months
* Systolic blood pressure > 150 or diastolic > 95 mm Hg
* Positive urine drug or alcohol screen
* Positive serology for HIV, HBV, or HCV
* History of alcoholism or drug abuse
* History of significant psychiatric disease, current depression of moderate or greater severity, any history of suicidal ideation
* Hypersensitivity to study drug or related compounds
* Use of prescription or OTC medication other than hormonal contraceptive within 14 days prior to first dosing with study drug
* Blood donation or significant blood loss within 56 days or plasma donation within 7 days prior to first dosing with study drug
* Women who are pregnant or lactating
* Hemoglobin < 12 g/dL
* Use of tobacco or nicotine-containing products within 6 months

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-07; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | One month

CONTACTS AND LOCATIONS:
Overall Officials: Wesley W Day, PhD, Study Director — VIVUS LLC
Locations (1):
- VIVUS, Inc., Mountain View, California, United States